CLINICAL TRIAL: NCT03208205
Title: Outcomes of Vitrectomy in Pediatric Retinal Detachment With Proliferative Vitreoretinopathy
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Other Study IDs: 0001
Record Dates: First submitted 2017-06-01; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Pediatric Rhegmatogenous Retinal Detachment
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: vitrectomy — Complete 23G PPV with scleral indentation was performed using Constellation system. Posterior vitreous detachment was induced very carefully by the cutter probe using aspiration. The peripheral vitreous was removed in all eyes with 360° of the vitreous base shaved under scleral indentation. After complete retinal attachment was achieved, endolaser photocoagulation was applied around the retinal break(s) as three to four rows of burns or/and cryopexy under HPFCL. Then a HPFCL/air/5000cst silicone oil exchange was performed. In one eye only HPFCL/air exchange was performed. Sclerotomies were sutured when needed with Vicryl 8.0 sutures.

SUMMARY:
The aim of this study is to report outcomes of pars plana vitrectomy (PPV) in pediatric retinal detachment (RD) accompanied with proliferative vitreoretinopathy (PVR) as well as complications and factors influencing the final anatomical and functional results.

This is retrospective consecutive case series of 14 eyes treated with primary PPV for RD repair. Average postoperative follow-up period is 34 months.

DETAILED DESCRIPTION:
This is the retrospective study of 14 consecutive patients younger than 18 years age who underwent primary PPV at the Department of General Ophthalmology of Medical University of Lublin in a time period from 1st January 2006 to 1st January 2017. This study followed the tenets of the Declaration of Helsinki. The treatment chosen in the study was a part of a standard care. Written informed consent was taken from all subjects. All patients underwent vitreoretinal surgery due to RD (rhegmatogenous, tractional or combined rhegmatogenous and tractional). Exclusion criteria from the study was the time of follow-up less than 6 months.

Average age at the time of the presence of RD was 10±4.7 years (range 4-17 years). Pre- and postoperative data were collected. Descriptive statistical analysis included gender, age at the presentation, laterality, etiology, duration of presenting symptoms, presences of ocular comorbidities, macular status (attached or non-attached), presence of PVR grade C, initial and final best-corrected visual acuity (BCVA), number of procedures, type of endotamponade during PPV, final lens status, duration of the follow-up, anatomical success and complications. Indications for PPV were as follows: presence of advanced PVR and/or total RD and/or multiple breaks, giant retinal tears. PVR was graded according to the Retina Society Terminology Classification [9]. Visual acuity was measured by Snellen charts. The anatomical success was defined as persistent retinal reattachment at the last follow-up visit (regardless of presence or absence of silicone oil tamponade).

Statistical computations were performed using STATISTICA 13PL (Stasoft, USA) programme.

ELIGIBILITY:
Inclusion Criteria:

* patients younger than 18 years age who underwent primary PPV at the Department of General Ophthalmology of Medical University of Lublin in a time period from 1st January 2006 to 1st January 2017

Exclusion Criteria:

* age up to 18 years old

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Persistent retinal reattachment | 30 months
  Pre- and postoperative data were collected. Descriptive statistical analysis included gender, age at the presentation, laterality, etiology, duration of presenting symptoms, presences of ocular comorbidities, macular status (attached or non-attached), presence of PVR grade C, initial and final best-corrected visual acuity (BCVA), number of procedures, type of endotamponade during PPV, final lens status, duration of the follow-up, anatomical success and complications. Indications for PPV were as follows: presence of advanced PVR and/or total RD and/or multiple breaks, giant retinal tears. PVR was graded according to the Retina Society Terminology Classification [9]. Visual acuity was measured by Snellen charts. The anatomical success was defined as persistent retinal reattachment at the last follow-up visit (regardless of presence or absence of silicone oil tamponade).
  Statistical computations were performed using STATISTICA 13PL (Stasoft, USA) programme

CONTACTS AND LOCATIONS:
Locations (1):
- General Department of Ophthalmology in Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Rejdak R, Nowakowska D, Wrona K, Maciejewski R, Junemann AG, Nowomiejska K. Outcomes of Vitrectomy in Pediatric Retinal Detachment with Proliferative Vitreoretinopathy. J Ophthalmol. 2017;2017:8109390. doi: 10.1155/2017/8109390. Epub 2017 Aug 3. PMID 28840039